CLINICAL TRIAL: NCT03938220
Title: Validation of Electrical Cardiometry Measurements Compared to Transthoracic Echocardiography in Fluid Responsiveness in Sepsis
Brief Title: Electrical Cardiometry Compared to Transthoracic Echocardiography in Fluid Responsiveness in Sepsis
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Assistant lecturer, Tanta University
Other Study IDs: 33017/03/19
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Electrical Cardiometry; Transthoracic Echocardiography; Fluid Responsiveness; Sepsis; Stoke Volume
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fluid responders: fluid responder if stroke volume increases by > 10% after the fluid challenge
  Interventions: Device: Electrical Cardiometry
- fluid non responders: fluid responder if stroke volume increases by <= 10% after the fluid challenge
  Interventions: Device: Electrical Cardiometry

INTERVENTIONS:
Device: Electrical Cardiometry — Electrical cardiometry (EC) measurements: by the ICON_ hemodynamic monitor (ICON Cardiotronics, Inc., La Jolla, CA 92307; Osyka Medical GmbH, Berlin, and Germany, model C3, Serial no: 1725303). Four sensors of EC will be applied (1st: 5 cm above the base of the neck, 2nd: on the base of neck, 3rd: lower thorax at the level of the xiphoid and 4th: 5 cm below the 3rd electrode at the level of anterior axillary line). The ICON continuously displays HR, SV and CO.

SUMMARY:
The aim of this study is to evaluate the diagnostic accuracy of electrical cardiometry (EC) for the noninvasive determination of fluid responsiveness in sepsis and agreement of (EC) compared to transthoracic echocardiography (TTE).

DETAILED DESCRIPTION:
Usual investigations [complete blood count (CBC), C reactive protein (CRP), serum procalcitonin, serum lactate, arterial blood gases (ABG), blood culture, electrocardiogram (ECG) and liver and renal function tests] will be done.

Once the diagnosis of sepsis is definite and the patient develops hypotension, all patients will undergo simultaneous measurement by (EC) using the ICON_ device and (TTE).

Electrical cardiometry (EC) measurements: by the ICON_ hemodynamic monitor (ICON Cardiotronics, Inc., La Jolla, CA 92307; Osyka Medical GmbH, Berlin, and Germany, model C3, Serial no: 1725303). Four sensors of (EC) will be applied (1st: 5 cm above the base of the neck, 2nd: on the base of the neck, 3rd: lower thorax at the level of the xiphoid and 4th: 5 cm below the 3rd electrode at the level of the anterior axillary line). The ICON continuously displays heart rate, stroke volume, and cardiac output.

Transthoracic echocardiography (TTE) measurements: will be performed by using Philips (CX50 - Extreme edition) equipped with echo probe. SV of the left ventricle will be calculated using LVOT diameter (D) just below the aortic valve from parasternal long-axis view and velocity time integral (VTI) measured in left ventricle outflow tract (LVOT) from apical 5 chamber view (by pulsed wave Doppler), respectively. The machine's built-in software uses the formula ''(πD2/4) × VTI × HR'' to calculate CO.

Management of sepsis will be done according to surviving sepsis campaign guidelines in 2016 and its update 2018.

Fluid resuscitation will be 30 mL/kg of intravenous infusion of lactated ringer to be given within the first 3 h (≈5 mL/kg/30 min) guided by fluid responsiveness (fluid responder if SV increases by > 10% after the fluid challenge). If the patient becomes fluid non-responder, vasopressor infusion (norepinephrine 0.05-0.3µg/kg/min) will start. The end of the study is when mean arterial blood pressure > 65 mmHg (either by fluid or both fluid and vasopressor).

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 65 years old.
* Clinical criteria of sepsis [acute change in sepsis-related organ failure assessment (SOFA) variables ≥ 2 points consequent to the infection which include: PaO2/FiO2 ratio < 300, Glasgow Coma Scale score < 15, mean arterial pressure (MAP) < 70 mmHg, serum creatinine >1.2 mg/dl or urine output < 0.5 ml/kg/h, serum bilirubin > 1.2 mg/dL, platelet count < 150 X 103 /µl].
* Developing hypotension (mean arterial blood pressure ≤ 65 mmHg).

Exclusion Criteria:

* Other causes of shock
* Previous cardiac disease
* Rhythm other than sinus rhythm or heart rate > 140 beats/min
* Chronic renal failure.

Ages: 19 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study will be carried out in Tanta University Hospitals at surgical ICU
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of electrical cardiometry to predict fluid responsiveness. | 24 hours
  Fluid resuscitation will be 30 mL/kg of intravenous infusion of lactated ringer to be given within the first 3 h (≈5 mL/kg/30 min) guided by fluid responsiveness (fluid responder if stroke volume increases by > 10% after the fluid challenge). If the patient becomes fluid non-responder, vasopressor infusion (norepinephrine 0.05-0.3µg/kg/min) will start. The end of the study is when mean arterial blood pressure> 65 mmHg (either by fluid or both fluid and vasopressor).

SECONDARY OUTCOMES:
Agreement of electrical cardiometry with transthoracic echocardiography in the change of stroke volume before and after fluid challenge. | 24 hours
  Fluid resuscitation will be 30 mL/kg of intravenous infusion of lactated ringer to be given within the first 3 h (≈5 mL/kg/30 min) guided by fluid responsiveness (fluid responder if stroke volume increases by > 10% after the fluid challenge). If the patient becomes fluid non-responder, vasopressor infusion (norepinephrine 0.05-0.3µg/kg/min) will start. The end of the study is when mean arterial blood pressure> 65 mmHg (either by fluid or both fluid and vasopressor).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt